CLINICAL TRIAL: NCT06953739
Title: A Multicenter, Randomized Controlled Clinical Study of Pegaspargase Combined With P-GEMD Regimen Versus P-Gemox Regimen in the Treatment of Untreated Early-Stage Non-Upper Aerodigestive Tract or Advanced-Stage Extranodal NK/T-Cell Lymphoma.
Brief Title: A Study Comparing of P-GEMD Regimen Versus P-Gemox Regimen With Untreated Early-Stage NUAT or Advanced-Stage ENKTL.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-NKTCL-K05
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: NK-T-Cell Lymphoma, Extranodal
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-GEMD (Experimental): The P-GEMD regimen (pegaspargase at 3750 IU, d2; gemcitabine at 1000 mg/m2, d1; etoposide at 65 mg/m2, d2-4; mitoxantrone hydrochloride liposome at 12mg/m2, d1; dexamethasone at 40 mg/d, d1-4.) was administered intravenously every 3 weeks until up to 6 cycles of planned therapy.
  Interventions: Drug: P-GEMD
- P-Gemox (Other): The P-Gemox regimen (pegaspargase at 2000-2500 IU/m2, d2; gemcitabine at 1000 mg/m2, d1, d8; oxaliplatin at 130 mg/m2, d1) was administered intravenously every 3 weeks until up to 6 cycles of planned therapy.
  Interventions: Drug: P-Gemox

INTERVENTIONS:
Drug: P-GEMD — Drug: Mitoxantrone hydrochloride liposome Mitoxantrone hydrochloride liposome (12 mg/m2) on day 1, every 3 weeks; Drug: Pegaspargase Pegaspargase(3750 IU) on day 2, every 3 weeks; Drug: Gemcitabine Gemcitabine (1000 mg/m2) on day 1, every 3 weeks; Drug: Etoposide Etoposide (65 mg/m2) on day 2-4, every 3 weeks. Drug: Dexamethasone Dexamethasone (40 mg/d) will be taken orally from day 1-4, every 3 weeks; Patients > 65 years of age may be adjusted according to the investigator's decision.
  Arms: P-GEMD
Drug: P-Gemox — Drug: Pegaspargase Pegaspargase(2000-2500 IU/m2) on day 1, every 3 weeks; Drug: Gemcitabine Gemcitabine (1000 mg/m2) on day 1 and day 8, every 3 weeks; Drug: Oxaliplatin Oxaliplatin (130mg/m2) on day 1, every 3 weeks; Patients > 65 years of age may be adjusted according to the investigator's decision.
  Arms: P-Gemox

SUMMARY:
Extranodal natural-killer (NK)/T-cell lymphoma (ENKTL) is an aggressive subtype of non-Hodgkin lymphoma with a poor prognosis. Notably, patients with advanced-stage disease or early-stage non-upper aero-digestive tract (NUAT) involvement frequently develop hemophagocytic lymphohistiocytosis (HLH), necessitating more effective therapeutic interventions. This Multicenter, Randomized Controlled Clinical Study aimed to compare the efficacy and safety of P-GEMD and P-Gemox in the treatment of newly diagnosed early NUAT or advanced-stage ENKTL.

DETAILED DESCRIPTION:
This Multicenter, Randomized Controlled Clinical Study aimed to compare the efficacy and safety of P-GEMD and P-Gemox in the treatment of newly diagnosed early NUAT or advanced-stage ENKTL. The P-GEMD regimen (pegaspargase; gemcitabine; etoposide; mitoxantrone hydrochlorid liposome; dexamethasone) was administered intravenously every 3 weeks until up to 6 cycles of planned therapy. The P-Gemox regimen ( Pegaspargase, Gemcitabine, and Oxaliplatin) was administered intravenously 3 weeks until up to 6 cycles of planned therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily join this study and sign the informed consent form; 2.Age ≥18 years old; 3.Expected survival time ≥ 3 months; 4. Histopathologically confirmed early non-upper aerodigestive or advanced ENKTL; 5. There must be at least one evaluable or measurable lesion that meets the Lugano2014 criteria: lymph node lesions, measurable lymph nodes need to have a long diameter > 1.5cm; non-lymph node lesions, extranodal lesions that can be measured Long diameter > 1.0cm; 6. ECOG score 0-2 points; 7. Bone marrow function: neutrophil count ≥ 1.5×109/L, platelet count ≥ 75×109/L, hemoglobin ≥ 80g/L(Restriction may be relaxed in patients with bone marrow involvement, Absolute neutrophil count (ANC) ≥1.0×109/L, Platelet count (PLT) ≥50×109/L, Hemoglobin(HB)≥ 75g/L); 8. Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of the normal value; alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 times the upper limit of the normal value (for patients with liver invasion ≤ 5 times the normal value upper limit); total bilirubin ≤ 1.5 times the upper limit of normal value (for patients with liver invasion ≤ 3 times the upper limit of normal value).

Exclusion Criteria:

* 1.Hypersensitivity to any study drug or its components; 2. Uncontrollable systemic diseases (such as advanced infection, uncontrollable hypertension, diabetes, etc.); 3. Cardiac function and disease meet one of the following conditions : A.long QTc syndrome or QTc interval >480 ms; B.complete left bundle branch block, second-degree or third-degree atrioventricular block; C.severe, uncontrolled arrhythmia requiring drug treatment ; D.New York Society of Cardiology ≥ Grade III; E.Cardiac ejection fraction (LVEF) lower than 50%; F.Myocardial infarction, unstable angina, and severely unstable ventricular rhythm within 6 months before recruitment History of arrhythmia or any other arrhythmia requiring treatment, history of clinically severe pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities.

  4. Active hepatitis B and C infection (positive hepatitis B virus surface antigen and more than 1x103 copies/mL of hepatitis B virus DNA; more than 1x103 copies/mL of hepatitis C virus RNA); 5. Human immunodeficiency virus (HIV) infection (positive HIV antibody); 6. Previously or currently suffering from other malignant tumors (except for effectively controlled non-melanoma skin basal cell carcinoma, breast/cervix carcinoma in situ and other malignant tumors that have been effectively controlled without treatment in the past five years); 7. Central nervous system (CNS) involvement at the time of recruitment; 8. Pregnant, lactating women and patients of childbearing age who do not want to take contraceptive measures; 9.Other investigators judge that they are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | 5.5years
  Response is assessed according to the lugano criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 5.5years
  Response is assessed according to the lugano criteria.
Progression-Free-Survival (PFS) | 5.5years
  From the time subjects were enrolled to the time of disease progression (in any way) or death from any cause.
Duration of Response (DOR) | 5.5years
  The time between meeting the criteria for treatment effectiveness (first recorded complete or partial response) and the first clear recurrence or progression.
Overall survival (OS) | 5.5years
  From the date of inclusion to date of death, irrespective of cause.
EBV-DNA load level (before and after treatment) | 5.5 years
  EBV-DNA was detected at time points before and after treatment.
Hematologic and non-hematologic toxicity. | From the first day of medication to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.Hematologic and non-hematologic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Principal Investigator — he First Affiliated Hospital with Nanjing Medical University, Nanjing, China; Jinhua Liang, Principal Investigator — he First Affiliated Hospital with Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No